CLINICAL TRIAL: NCT00898053
Title: Observational - Prognostic Value of p53 and/or p16 Alterations in Ewing Sarcoma
Brief Title: Study of Tumor Samples From Patients With Ewing Sarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEWS08B1; NCI-2009-00372 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA098543 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Localized Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Previously archived tumor samples are analyzed for p53 mutations and p16 deletion by immunohistochemistry, FISH, PCR, and DNA sequencing.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is looking at tumor samples from patients with Ewing sarcoma. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Prospective Biospecimen Retention: Samples With DNA Biospecimen Description: Tissue Study Population Description: Samples collected from AEWS0031 and patients registered on AEWS08B1 Sampling Method: Non-Probability Sample

PRIMARY OBJECTIVES:

I. Determine if mutation of p53, and/or deletion of the p16 locus, have prognostic value in patients with Ewing sarcoma.

SECONDARY OBJECTIVES:

I. Estimate the incidence of p53 mutation in Ewing sarcoma samples collected from COG studies.

II. Estimate the incidence of p16 deletions in Ewing sarcoma samples collected from COG studies.

III. Prepare and archive amplified genomic DNA from Ewing sarcoma samples collected from COG studies for future biologic analysis.

OUTLINE: This is a multicenter study.

Previously archived tumor samples are analyzed for p53 mutations and p16 deletion by immunohistochemistry, FISH, PCR, and DNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ewing sarcoma
* Banked specimens from patients enrolled on AEWS0031

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of Ewing sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Event-free survival | Time from study entry until disease progression, death without progression of disease, occurrence of a second malignant neoplasm or last follow-up, assessed up to 3 years

SECONDARY OUTCOMES:
Incidence of p53 mutations using the model of Sather and Sposto | Baseline
  Assessed using a two sided log rank test. The expected 95% confidence interval associated with this estimate, as a function of sample size and true mutation/deletion frequency is provided.
Incidence of p16 loss or deletion using the model of Sather and Sposto | Baseline
  Assessed using a two sided log rank test. The expected 95% confidence interval associated with this estimate, as a function of sample size and true mutation/deletion frequency is provided.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lessnick, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States